CLINICAL TRIAL: NCT03224598
Title: A Phase 2 Open Label Study of A-101 Topical Solution in Subjects With Dermatosis Papulosa Nigra
Brief Title: A Study of A-101 Topical Solution in Subjects With Dermatosis Papulosa Nigra
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-101-DPN-201
Record Dates: First submitted 2017-07-05; First posted 2017-07-21 (Actual); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-02

CONDITIONS: Dermatosis Papulosa Nigra
MeSH Terms: conditions — Dermatosis Papulosa Nigra

STUDY DESIGN:
Intervention Model Description: The first cohort of the study will enroll a total of 12 subjects. In the second part of the study, subjects will be a randomized to additional two-arm cohorts. Subjects will be randomized to one of the following 2 treatment arms:
  * A-101 40% without medically abrading the identified DPN prior to treatment
  * A-101 40% with the identified DPN lesions medically abraded prior to treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- No medical abrading (Experimental): A-101 40% without medically abrading the identified DPN prior to treatment
  Interventions: Drug: A-101 Topical Solution 40%
- Medically abrading (Experimental): A-101 40% with the identified DPN lesions medically abraded prior to treatment
  Interventions: Drug: A-101 Topical Solution 40%
- Initial cohort - no medical abrading (Experimental): A-101 40% without medically abrading the identified DPN prior to treatment
  Interventions: Drug: A-101 Topical Solution 40%

INTERVENTIONS:
Drug: A-101 Topical Solution 40% — A-101 Topical Solution 40%

SUMMARY:
Evaluate the safety and efficacy of hydrogen peroxide, A-101 Solution 40% for the treatment of DPN lesions on subjects with a Fitzpatrick Skin Type of 5 or 6.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the safety and efficacy of hydrogen peroxide, A-101 Solution 40% for the treatment of DPN lesions on subjects with a Fitzpatrick Skin Type of 5 or 6.

The secondary objectives of this study include:

* Durability of response
* Safety

An exploratory objective of this study will evaluate the subject's assessment of the treatment of A-101 to DPN lesions using a Subject Self-Assessment Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Provisions of written informed consent for participation in this study.
2. Male or female ≥ 18 years old.
3. Subject has a clinical diagnosis of dermatosis papulose nigra.
4. Fitzpatrick Skin Type of 5 or 6
5. Subject has 4 target DPN lesions located in an area that has not been previously treated.
6. Subject chemistry and complete blood count results are within normal limits for the central laboratory.
7. Woman of childbearing potential must have a negative urine pregnancy test within 14 days of the first application of study drug and agree to use an active method of birth control for the duration of the study
8. Subject is non-pregnant and non-lactating.
9. Subject is in good general health and free of any known disease state or physical condition.
10. Subject is willing and able to follow all study instructions and to attend all study visits.

Exclusion Criteria:

1. Subject has clinically atypical and /or rapidly growing DPN lesion.
2. Subject has current systemic malignancy.
3. Subject has a history of keloids
4. Subject has a history of post inflammatory hyperpigmentation lasting longer than 1 year.
5. Subject has used any of the following systemic therapies within the specified period prior to Visit 1:

   * Retinoids; 180 days
   * Corticosteroids; 28 days
   * Antimetabolites (e.g., methotrexate); 28 days
6. Subject has used any of the following topical therapies within the specified period prior to Visit 1 on, or in a proximity to any Target Lesion, that in the investigator's opinion interferes with the study medication treatment or the study assessments:

   * LASER, light or other energy based therapy (e.g., intense pulsed light [IPL], photo-dynamic therapy [PDT]; 180 days
   * Liquid nitrogen, electrodesiccation, curettage, imiquimod, 5-fluoruracil (5FU), or ingenol mebutate; 60 days
   * Retinoids; 28 days
   * Microdermabrasion or superficial chemical peels; 14 days
   * Corticosteroids or antibiotics; 14 days.
7. Subject currently has or has had any of the following within the specified period prior to Visit 1 on or in a proximity to any Target Lesion that, in the investigator's opinion, interferes with the study medication treatment or the study assessments:

   * Cutaneous malignancy; 180 days
   * Sunburn; currently
   * Pre-malignancy (e.g. actinic keratosis); currently
   * Body art (e.g. tattoos, piercing, etc.); currently
   * Excessive tan. The use of self-tanning lotions/sprays are prohibited.
8. Subject has a history of sensitivity to any of the ingredients in the study medications.
9. Subject has any current skin disease (e.g. psoriasis, atopic dermatitis, eczema, sun damage), or condition (e.g. sunburn, excessive hair, open wounds) that, in the opinion of the investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations.
10. Participation in another therapeutic investigational drug trial in which administration of an investigational study medication occurred with 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Aclaris Investigational Site, Washington D.C., District of Columbia
  - Aclaris Investigational Site, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Initial Cohort - no Medical Abrading: initial cohort no medical abrading different treatment schedule
Period: Overall Study
Arm/Group | No Medical Abrading | Medically Abrading | Initial Cohort - no Medical Abrading
Started | 9 | 17 | 13
Completed | 9 | 14 | 13
Not Completed | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Medical Abrading | Medically Abrading | Initial Cohort - no Medical Abrading | Total
Number analyzed (Participants) | 9 | 17 | 13 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 11 | 6 | 22
  >=65 years | 4 | 6 | 7 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 8 | 29
  Male | 1 | 4 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 16 | 13 | 38
  White | 0 | 1 | 0 | 1
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 17 | 13 | 39
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  fitzpatrick 5: Rarely burns, tans darkly easily | 7 | 10 | 8 | 25
  fitzpatrick 6: Never burns, always tans darkly | 2 | 7 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Physician's DPN Lesions Assessment
Description: Efficacy endpoints will include summary statistics (frequency distributions, proportions, means, medians and standard deviations, as appropriate) by visit for the following parameters: Physician's DPN Lesion Assessment scale results per treated lesion, subject responders defined by Physician's DPN Lesion Assessment scale outcome, and changes from baseline treated lesion diameter
  Physician's DPN Lesion Assessment Grade Descriptor 0 Clear: no visible DPN lesion;
  1. Near Clear: a slightly visible DPN lesion; lesion may be macular
  2. Small: a visible DPN lesion with a diameter of less than 3 mm
  3. Large : a visible DPN lesion that is elevated with a diameter of ≥3 mm
Time Frame: Day 106
Population: per-protocol
Measure: Mean (Standard Deviation); unit: score on a scale (PLA)
Arm/Group | No Medical Abrading | Medically Abrading | Initial Cohort - no Medical Abrading
Number analyzed (Participants) | 9 | 14 | 13
score on a scale (PLA) | -0.75 (0.52) | -1.38 (0.90) | -0.92 (0.95)

ADVERSE EVENTS:
Time Frame: 106 days
Description: An adverse event (AE) is any untoward medical occurrence in a patient that develops or worsens in severity during the conduct of a clinical study of a pharmaceutical product and does not necessarily have a causal relationship to the study drug.
  assessed at all visits
Arm/Group | No Medical Abrading | Medically Abrading | Initial Cohort - no Medical Abrading
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/17 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 1/9 | 2/17 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Medical Abrading (N=9) | Medically Abrading (N=17) | Initial Cohort - no Medical Abrading (N=13)
eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT03224598/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT03224598/SAP_001.pdf